CLINICAL TRIAL: NCT04842916
Title: InteGRAtive Analysis of TuMor, Microenvironment, ImmunitY and Patient Expectation for Personalized Response Prediction in Gastric Cancer
Acronym: GRAMMY
Status: Recruiting | Type: Observational
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Collaborators: ERA PERMED (Unknown)
Responsible Party: Sponsor
Other Study IDs: IRSTB111
Record Dates: First submitted 2020-12-23; First posted 2021-04-13 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Gastric Cancer
Keywords: Gastric cancer, Chemotherapy, Response, Personalized medicine
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Formalin Fixed Paraffin Embedded (FFPE) tissue, Blood, Fresh Frozen (FF) tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Gastric cancer patients: gastric cancer patients with histologically confirmed, potentially resectable adenocarcinoma of the stomach or the gastroesophageal junction receiving the standard of medical care in Europe

SUMMARY:
Multicentric, exploratory, non-pharmacologic, retrospective/prospective, translational study aiming to identify the molecular, cellular and psychological-sociological variables predictive of response to chemotherapy in gastric cancer patients.

DETAILED DESCRIPTION:
Gastric cancer (GC) is a complex disease that represents the fifth most common malignancy in the world and the third leading cause of cancer death in both sexes. Chemotherapy (CT) combined with surgery represents the standard of care for stages II-III GC, but the efficacy of such treatments is still limited for many patients. It is mandatory to develop novel strategies aimed at identifying predictive markers, as well as deciphering the impact of the psychological-social and cultural environment of each patient on the outcome. GRAMMY study proposes a novel interdisciplinary approach integrating high impact basic, translational and psychological/sociological research towards developing an optimized patient stratification tool for the early prediction of therapy-resistant GC patient groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of histologically confirmed, potentially resectable adenocarcinoma of the stomach (GC) or the gastric-esophageal junction (GEJ) treated with the standard regimens (5-Fluoro-Uracil or Capecitabine + Oxaliplatin +/- Docetaxel)
* Participant is willing and able to give informed consent for participation in the study (prospective and retrospective cohort) or Substitutive Informed Consent Declaration Form will be subscribed by the PI for patients that are not reachable
* Male or Female, aged >18 years
* Availability of tissue samples and clinico-pathological data for retrospective cohort

Exclusion Criteria:

* Age < 18 years
* Early Gastric Cancer and T2 (if N0)
* Linitis plastica
* Positive peritoneal cytology or peritoneal involvement
* Distant metastases
* Patient refusal to participate
* Patient refusal to the use of their own samples for research
* Patient withdrawing from treatment plan whilst under therapy due to patient co-morbidities or failure to comply with clinical counselling
* Patients with underlying pathologies rendering sampling of biological material either as endangering patient's clinical status or as unusable
* Patients with mental illness hindering the capacity to provide precise information in questionnaires or successfully comply with caregiver's recommendations

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with potentially resectable adenocarcinoma of the stomach (GC) or the gastric-esophageal junction (GEJ) who received pre- or peri-operative chemotherapy or up-front surgery followed by chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-09-22 (Actual); Primary Completion 2027-05-22 (Estimated); Study Completion 2027-05-22 (Estimated)

PRIMARY OUTCOMES:
Genomic alterations in tumoral tissue in responders and non-responders | 36 months
  Number of Genomic alterations in tumoral tissue
Quantitative and qualitative analysis of the tumor microenvironment composition in responders and non-responders | 36 months
  Analysis of type and size of immune cell subpopulations surrounding primary tumor and extracellular matrix composition on FFPE samples collected at diagnosis and/or surgery. Correlation of data acquired to Participant's response score (TRG or DFS).
Analysis of cell-free DNA (cfDNA) from blood samples in responders and non-responders | 36 months
  cfDNA will be quantified in Participant's peripheral blood derivatives (plasma, serum) and characterized for Genomic alterations. Samples will be obtained (1) prior to and (2) by completion of chemotherapy in the Neoadjuvant Chemotherapy (NCT) treated cohorts, together with sampling after surgery (3). TRG score will be utilized as measure of response. Accordingly, in NCT-naive cohorts, analysis of samples obtained 1) pre- operatively and 2) by completion of post-operative chemotherapy treatment will be correlated with the respective Disease-Progression clinical indicators.
Analysis of circulating tumor cells (CTC) from blood samples in responders and non-responders. | 36 months
  gene expression profile of CTC cells (when isolated in sufficient quantity)
Peripheral blood mononuclear cells (PBMCs) and host immunity parameters in responders and non-responders | 36 months
  Phenotype analysis of representative immune cell subpopulations (i.e. monocytes, helper T cells, cytotoxic T cells, Tregs, Natural Killer (NK) /NKT) in Participants' peripheral blood samples obtained prior- and post- treatment. Combinational analysis of data acquired in correlation with Patient's response score.

SECONDARY OUTCOMES:
Psychological status of patients in relation to therapy response | 36 months
  Psychological status of patients in relation to therapy response evaluated by a psychologist through structured interview

CONTACTS AND LOCATIONS:
Overall Officials: Chiara Molinari, Study Chair — IRST IRCCS
Locations (5):
- France (2):
  - Centre Hospitalier Regional et Universitaire (CHRU), Brest
  - INSERM, Faculty of Medicine (UMR1078), Brest
- 1st Department of Propaedeutic Surgery, National & Kapodistrian University of Athens (NKUA), Athens, Greece
- Italy (2):
  - IRST IRCCS UO Oncologia, Meldola
  - AUSL Romagna, UO Oncologia, Ravenna